CLINICAL TRIAL: NCT04295824
Title: Skin Pathology Assessment With Optical Technologies (SPOT): a Cross- Sectional Clinical Study in Atopic Dermatitis Patients and Healthy Subjects
Brief Title: Skin Pathology Assessment With Optical Technologies
Acronym: SPOT
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20628
Record Dates: First submitted 2020-02-25; First posted 2020-03-05 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Atopic Dermatitis Eczema
Keywords: atopic dermatitis; atopic eczema; optical coherence tomography; skin biopsy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva sample (buccal swab) for FLG genotyping. Superficial stratum corneum sample collection by tape-stripping: For determination of protease activity ex vivo and determination of natural moisturizing factor (NMF) levels by HPLC. FibroTX SELF samples will be collected from the designated skin sites using a transdermal patch system to collect secreted and diffusible regulatory molecules directly from the skin surface according to the manufacturer's instructions. Using this system multiple analytes can be measured, including for example CXCL1, IL-1A, CCL27, and hBD2. Blood samples will be collected for future study of cytokine levels in relationship to the structural changes observed within the skin. Skin Biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild AD: 20 subjects with mild local AD on their volar forearm (At least 10 with lesions on the face | At least 10 which are globally mild).
  Interventions: Diagnostic Test: Skin imaging and Skin biopsy
- Moderate AD: 20 subjects with moderate local AD on their volar forearm (At least 10 with lesions on the face | At least 10 which are globally moderate).
  Interventions: Diagnostic Test: Skin imaging and Skin biopsy
- Severe AD: 20 subjects with severe local AD on their volar forearm (At least 10 with lesions on the face | At least 10 which are globally severe).
  Interventions: Diagnostic Test: Skin imaging and Skin biopsy
- Healthy: 20 healthy volunteers
  Interventions: Diagnostic Test: Skin imaging and Skin biopsy

INTERVENTIONS:
Diagnostic Test: Skin imaging and Skin biopsy — Imaging includes:
  * Structural Optical Coherence Tomography (OCT) - Skin thickness/roughness.
  * Angiographic OCT- Vessel depth/morphology.
  * Polarisation-sensitive OCT - Tissue birefringence / collagen index.
  * Skin biopsies will be taken from the same volar forearm site as the imaging is performed.

SUMMARY:
The Skin Pathology assessment with Optical Technologies (SPOT) study aims to assess the feasibility of recently developed light-based skin imaging tools such as Optical Coherence Tomography (OCT) for the study of eczema (dermatitis [AD]).

Tools such as OCT have enabled us to see beneath the skin surface, allowing us to see changes in our skin which are hidden and impossible to assess by eye, simply by shining harmless light into the skin. The investigators want to understand what these changes represent in the broader context of eczema.

To do this, the investigators would like to recruit 60 volunteers who have a range of different eczema severities. The investigators would also like to recruit 20 healthy volunteers, who have never suffered from eczema. All volunteers would be aged between 11 and 60.

The study is based at the Royal Hallamshire Hospital in Sheffield, with consent and sample-collection taking place at either the hospital's Clinical Research Facility or the Sheffield Children's Hospital. The study consists of a single main visit, which is expected to take approximately 3 hours, and a short follow up visit 2-4 weeks later.

During the main study visit, the investigators will collect a range of measurements from the inner elbows and cheeks using harmless topical probes (Including OCT). These measurements include information about the skin's layers, blood flow, composition, water loss, acidity and redness. The investigators will also collect some samples, including tape-strips, a saliva sample and blood samples. For adult participants the investigators will also collect 2-4 skin biopsies from the inner elbows, which involves removing small pieces of skin under a local anaesthetic.

It is our hope that by demonstrating the advantages of new harmless imaging techniques, the investigators can reduce the need for invasive procedures in the future. Long term, this may help us to improve the way healthcare professionals monitor and treat eczema.

DETAILED DESCRIPTION:
A total of 80 participants will be recruited for the study spread equally across 4 cohorts, those with healthy skin, and those with a mild/moderate/severe eczema/dermatitis [AD] lesion on their inner elbow.

Our first point of contact with the participant involves providing them with a copy of the age-appropriate PIS and completing an expression of interest (EOI) form through phone/email/post. The EOI form contains questions for pre- screening purposes so that the likelihood of suitability can be estimated in order to avoid wasting the time of people who clearly don't meet the basic entry criteria (severity will need to be assessed during the screening visit). For volunteers who meet the basic entry criteria as outlined on the EOI form, the investigators will make it clear that the next step will be for a researcher on our team to contact them to arrange a screening/informed consent session at our test facility.

A member of the team will then contact interested volunteers to arrange their visit, at least 24 hours following the provision of the PIS. The bulk of the study consists of a single visit, which contains the full screening process, informed consent and the study protocol (A second short follow up visit 2-3 weeks later is also required for those providing biopsies).

When the participant arrives at either the Sheffield Children's Hospital (For adolescents) or the Royal Hallamshire Hospital Clinical Research Facility (Adults), a nurse will talk the participant through the study and what it involves. They will also be asked some basic questions about their skin and current medication. Their skin will be inspected visually by eye to assess eligibility and cohort allocation. If the participant is eligible, then they will be required to fill in an informed consent form (11-15 year olds will complete an assent form, with their legal guardian completing a consent form).

Following consent, the participants will be taken to the Royal Hallamshire Hospital Skin Research room. They will be asked to roll up their sleeves such that their elbows are able to acclimatise for 20 minutes. While waiting, the scan sites will be marked on the participants elbows using a washable ink (Scan sites on the cheeks will not be marked with ink) and a skin questionnaire will be conducted which asks basic questions about the history of eczema at each scan site. When ready, images will be collected from the scan sites using handheld probes which gently contact the skin surface. All of the images collected are completely harmless, and simply involve shining light into the skin. The following measurements will be collected in order: Clinical Photographs (From elbows and cheeks), Trans-epidermal water loss measurements (From elbows and cheeks), skin redness (From elbows and cheeks), FTIR spectra (From elbows and cheeks), Optical Coherence Tomography (From elbows and cheeks), Laser doppler images (From elbows), Polarisation-sensitive Optical Coherence Tomography (From elbows) and skin pH (From elbows and cheeks).

Once the images are collected, some samples will be collected from the participant. These include a buccal (Saliva) sample collected from the cheek and tape-strip/FIBROTX samples collected from the elbows. Both of the latter sampling methods involve sticking a patch onto the skin and gently peeling it off, which collects just the molecules/cells at the surface of the skin.

Following this sample collection, the participants will be taken back to the Sheffield Children's Hospital (For adolescents) or the Royal Hallamshire Hospital Clinical Research Facility (Adults) and a total of three 5ml blood samples will be collected from their arm. Adult participants will be required to provide at least 2 biopsies from their elbow at this point, this involves small pieces of skin being removed under local anaesthetic so that they can be viewed under a microscope. A further 2 biopsies are optional depending on consent.

As mentioned above, participants that provided biopsies will be required to attend a follow-up visit 2-4 weeks later in order to remove any stitches and check the health of the biopsy site.

All research data collected in the pursuit of this study, will be collected in pseudo-anonymised form. For the purposes of this study, "pseudo-anonymised research data" is data that has had all personal identifiable information (such as name, initials and date of birth) replaced by the subject identifier (unique study number), and so protects the identities on the participants whilst still enabling the information to be traced back by the direct study team (who will have access to the study number allocation).

Following the study visit, the pseudo-anonymised electronic data will be stored on a secure Sheffield Corporate Information and Computing Services (CICS) managed server with access limited to study delegates only. Any paper records will be stored in locked cabinets in the study rooms/offices. Patch samples will be sent to FIBROTX for analysis - any remaining samples will be sent to a biobank where consent has been explicitly provided. The two required biopsies will be gifted to Leo Pharma who will undertake study specific analysis, any remaining tissue will be entered into a biobank hosted by BioStorage Technologies GmbH on behalf of Leo Pharma. The optional biopsies will be analysed by researchers at the University of Sheffield, any remaining tissue will be entered into the University Of Sheffield Biobank so that it can be made available for use on future research studies. The first blood sample will be processed by Laboratory Medicine at the Northern General Hospital in Sheffield, the second will be gifted to Leo Pharma, and stored in a biobank hosted by BioStorage Technologies GmbH where it will be available to LEO Pharma and their research partners, the third will be stored in the University of Sheffield Biobank. Extracted DNA (from the saliva samples) will be kept for a maximum of 10 years by the University of Sheffield in the care of the Principal Investigator, so that it may be used to support future genetic studies.

Electronic data from the study will be analysed at Sheffield following the study completion. Information from this study will be used to write scientific reports and publications, but they will not include any information which makes it possible for participants to be identified. A summary of findings will be distributed to all participants at the close of the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects and AD patients

1. Male or female
2. Aged between 11-60 years
3. Volunteer understands the purpose, modalities and potential risk of the trial
4. Volunteers able to read and understand English
5. Volunteers willing to sign the informed consent

AD patients:

1. Volunteers with AD defined according to the UK working party diagnostic criteria
2. Must have an AD lesion present at either the right or left forearm (Proximal end).
3. For 10 participants in each AD group: visible AD lesion present on either the right or left cheek.
4. For 10 participants in each AD group: Global severity score (EASI) that matches their cohort allocation (Mild/Moderate/Severe).

According to the UK working party diagnostic criteria, eczema is defined as exhibiting an itchy skin condition plus 3 or more of:

* History of involvement of the skin creases
* Personal history of asthma or hay fever
* History of generally dry skin in past year
* Visible flexural dermatitis
* Onset below age 2

Instructions to participants 1. Do not ingest caffeine (e.g Coffee) or take anti-inflammatory drugs (e.g Ibuprofen) on the imaging day (until after imaging).

Exclusion Criteria:

1. Treatment with the following medications within 4 weeks: systemic immunosuppressive/immunomodulating drugs (e.g. methotrexate, cyclosporine, azathioprine, mycophenolate-mofetil, Janus kinase inhibitors, etc.), systemic corticosteroids.
2. Three or more bleach baths during any week within 4 weeks.
3. Treatment with biologics within 5 half-lives (if known) or 12 weeks.
4. Treatment with the following medications within 2 weeks if mild/moderate global severity or 1 week if severe global severity: topical corticosteroids, topical calcineurin inhibitors.
5. Treatment with any topical leave-on product on the test areas 7 days prior to participation if healthy/mild and 24 hours prior to participation if moderate/severe global severity.
6. Volunteers with acne, suntan, birth marks, multiple nevi, tattoos, blemishes or dense body hair that obstruct the test areas.
7. Volunteers with a condition that in the opinion of the investigator contradicts participation in the study.
8. Volunteer is incapable of giving fully informed consent.
9. Volunteers judged by the PI to be inappropriate for the trial.

Ages: 11 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient with atopic dermatitis/atopic eczema and Healthy Controls
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Local clinical severity | baseline visit 1
  Primary endpoint: Local clinical severity (erythema, papulation, excoriation and lichenification) of test skin sites

SECONDARY OUTCOMES:
Skin epidermal thickness | baseline visit 1
  Inflammation associated endpoint using Vivosight OCT system
Skin vascular plexus depth | baseline visit 1
  Inflammation associated endpoint using Vivosight OCT system
Skin vascular density/diameter | baseline visit 1
  Inflammation associated endpoint using Vivosight OCT system
Skin collagen index | baseline visit 1
  Inflammation associated endpoint using PS-OCT system
Skin surface roughness | baseline visit 1
  Inflammation associated endpoint using Vivosight OCT system
Epidermal layer scattering | baseline visit 1
  Inflammation associated endpoint putatively relating to tissue remodelling using Vivosight OCT system
Erythema index | baseline visit 1
  Inflammation associated endpoint using c-cube images of skin lesions
Stratum corneum structure | baseline visit 1
  Skin barrier associated endpoint using (ATR-FTIR) spectroscopy
Protease activity | baseline visit 1
  Skin barrier associated endpoint, Ex vivo, using superficial stratum corneum samples collected on D-Squame tape discs

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cork, MD+PhD, Principal Investigator — University of Sheffield & Sheffield Teaching Hospitals; Simon G Danby, PhD, Study Chair — University of Sheffield
Locations (1):
- Sheffield Dermatology Research, University of Sheffield Medical School, The Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverberg JI, Hanifin JM. Adult eczema prevalence and associations with asthma and other health and demographic factors: a US population-based study. J Allergy Clin Immunol. 2013 Nov;132(5):1132-8. doi: 10.1016/j.jaci.2013.08.031. Epub 2013 Oct 4. PMID 24094544
- [Background] Odhiambo JA, Williams HC, Clayton TO, Robertson CF, Asher MI; ISAAC Phase Three Study Group. Global variations in prevalence of eczema symptoms in children from ISAAC Phase Three. J Allergy Clin Immunol. 2009 Dec;124(6):1251-8.e23. doi: 10.1016/j.jaci.2009.10.009. PMID 20004783
- [Background] Holgate ST. The epidemic of allergy and asthma. Nature. 1999 Nov 25;402(6760 Suppl):B2-4. doi: 10.1038/35037000. PMID 10586888
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575
- [Background] Tang TS, Bieber T, Williams HC. Are the concepts of induction of remission and treatment of subclinical inflammation in atopic dermatitis clinically useful? J Allergy Clin Immunol. 2014 Jun;133(6):1615-25.e1. doi: 10.1016/j.jaci.2013.12.1079. Epub 2014 Mar 18. PMID 24655575
- [Background] Gfesser M, Abeck D, Rugemer J, Schreiner V, Stab F, Disch R, Ring J. The early phase of epidermal barrier regeneration is faster in patients with atopic eczema. Dermatology. 1997;195(4):332-6. doi: 10.1159/000245983. PMID 9529552
- [Background] Seidenari S, Giusti G. Objective assessment of the skin of children affected by atopic dermatitis: a study of pH, capacitance and TEWL in eczematous and clinically uninvolved skin. Acta Derm Venereol. 1995 Nov;75(6):429-33. doi: 10.2340/0001555575429433. PMID 8651017
- [Background] Kelleher M, Dunn-Galvin A, Hourihane JO, Murray D, Campbell LE, McLean WHI, Irvine AD. Skin barrier dysfunction measured by transepidermal water loss at 2 days and 2 months predates and predicts atopic dermatitis at 1 year. J Allergy Clin Immunol. 2015 Apr;135(4):930-935.e1. doi: 10.1016/j.jaci.2014.12.013. Epub 2015 Jan 22. PMID 25618747 (Retraction: PMID 33832697 J Allergy Clin Immunol. 2021 Apr;147(4):1526)
- [Background] Eberlein-Konig B, Spiegl A, Przybilla B. Change of skin roughness due to lowering air humidity in climate chamber. Acta Derm Venereol. 1996 Nov;76(6):447-9. doi: 10.2340/0001555576447449. PMID 8982408
- [Background] Eberlein-Konig B, Schafer T, Huss-Marp J, Darsow U, Mohrenschlager M, Herbert O, Abeck D, Kramer U, Behrendt H, Ring J. Skin surface pH, stratum corneum hydration, trans-epidermal water loss and skin roughness related to atopic eczema and skin dryness in a population of primary school children. Acta Derm Venereol. 2000 May;80(3):188-91. doi: 10.1080/000155500750042943. PMID 10954209
- [Background] Knor T, Meholjic-Fetahovic A, Mehmedagic A. Stratum corneum hydration and skin surface pH in patients with atopic dermatitis. Acta Dermatovenerol Croat. 2011;19(4):242-7. PMID 22185924
- [Background] Linde YW. Dry skin in atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1992;177:9-13. PMID 1466189
- [Background] Imokawa G. A possible mechanism underlying the ceramide deficiency in atopic dermatitis: expression of a deacylase enzyme that cleaves the N-acyl linkage of sphingomyelin and glucosylceramide. J Dermatol Sci. 2009 Jul;55(1):1-9. doi: 10.1016/j.jdermsci.2009.04.006. Epub 2009 May 13. PMID 19443184
- [Background] van Neste D, Douka M, Rahier J, Staquet MJ. Epidermal changes in atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1985;114:67-71. doi: 10.2340/000155551146771. PMID 3859169
- [Background] Byers RA, Maiti R, Danby SG, Pang EJ, Mitchell B, Carre MJ, Lewis R, Cork MJ, Matcher SJ. Sub-clinical assessment of atopic dermatitis severity using angiographic optical coherence tomography. Biomed Opt Express. 2018 Mar 29;9(4):2001-2017. doi: 10.1364/BOE.9.002001. eCollection 2018 Apr 1. PMID 29675335
- [Background] Cossmann M, Welzel J. Evaluation of the atrophogenic potential of different glucocorticoids using optical coherence tomography, 20-MHz ultrasound and profilometry; a double-blind, placebo-controlled trial. Br J Dermatol. 2006 Oct;155(4):700-6. doi: 10.1111/j.1365-2133.2006.07369.x. PMID 16965418
- [Background] Josse G, Rouvrais C, Mas A, Haftek M, Delalleau A, Ferraq Y, Ossant F, George J, Lagarde JM, Schmitt AM. A multitechnique evaluation of topical corticosteroid treatment. Skin Res Technol. 2009 Feb;15(1):35-9. doi: 10.1111/j.1600-0846.2008.00326.x. PMID 19152576
- [Background] Oh MH, Oh SY, Yu J, Myers AC, Leonard WJ, Liu YJ, Zhu Z, Zheng T. IL-13 induces skin fibrosis in atopic dermatitis by thymic stromal lymphopoietin. J Immunol. 2011 Jun 15;186(12):7232-42. doi: 10.4049/jimmunol.1100504. Epub 2011 May 16. PMID 21576506
- [Background] Welzel J, Lankenau E, Birngruber R, Engelhardt R. Optical coherence tomography of the human skin. J Am Acad Dermatol. 1997 Dec;37(6):958-63. doi: 10.1016/s0190-9622(97)70072-0. PMID 9418764
- [Background] Israelsen NM, Maria M, Mogensen M, Bojesen S, Jensen M, Haedersdal M, Podoleanu A, Bang O. The value of ultrahigh resolution OCT in dermatology - delineating the dermo-epidermal junction, capillaries in the dermal papillae and vellus hairs. Biomed Opt Express. 2018 Apr 19;9(5):2240-2265. doi: 10.1364/BOE.9.002240. eCollection 2018 May 1. PMID 29760984
- [Background] Maiti R, Gerhardt LC, Lee ZS, Byers RA, Woods D, Sanz-Herrera JA, Franklin SE, Lewis R, Matcher SJ, Carre MJ. In vivo measurement of skin surface strain and sub-surface layer deformation induced by natural tissue stretching. J Mech Behav Biomed Mater. 2016 Sep;62:556-569. doi: 10.1016/j.jmbbm.2016.05.035. Epub 2016 Jun 5. PMID 27310571
- [Background] Barton J, Stromski S. Flow measurement without phase information in optical coherence tomography images. Opt Express. 2005 Jul 11;13(14):5234-9. doi: 10.1364/opex.13.005234. PMID 19498514
- [Background] Chen CL, Wang RK. Optical coherence tomography based angiography [Invited]. Biomed Opt Express. 2017 Jan 24;8(2):1056-1082. doi: 10.1364/BOE.8.001056. eCollection 2017 Feb 1. PMID 28271003
- [Background] de Boer JF, Hitzenberger CK, Yasuno Y. Polarization sensitive optical coherence tomography - a review [Invited]. Biomed Opt Express. 2017 Feb 24;8(3):1838-1873. doi: 10.1364/BOE.8.001838. eCollection 2017 Mar 1. PMID 28663869
- [Background] Chopra R, Vakharia PP, Sacotte R, Patel N, Immaneni S, White T, Kantor R, Hsu DY, Silverberg JI. Severity strata for Eczema Area and Severity Index (EASI), modified EASI, Scoring Atopic Dermatitis (SCORAD), objective SCORAD, Atopic Dermatitis Severity Index and body surface area in adolescents and adults with atopic dermatitis. Br J Dermatol. 2017 Nov;177(5):1316-1321. doi: 10.1111/bjd.15641. Epub 2017 Oct 1. PMID 28485036
- [Background] Williams HC. Diagnostic criteria for atopic dermatitis. Lancet. 1996 Nov 16;348(9038):1391-2. doi: 10.1016/S0140-6736(05)65466-9. No abstract available. PMID 8918311
- [Background] Emerson RM, Charman CR, Williams HC. The Nottingham Eczema Severity Score: preliminary refinement of the Rajka and Langeland grading. Br J Dermatol. 2000 Feb;142(2):288-97. doi: 10.1046/j.1365-2133.2000.03300.x. PMID 10730763
- [Background] Imhof RE, De Jesus ME, Xiao P, Ciortea LI, Berg EP. Closed-chamber transepidermal water loss measurement: microclimate, calibration and performance. Int J Cosmet Sci. 2009 Apr;31(2):97-118. doi: 10.1111/j.1468-2494.2008.00476.x. Epub 2009 Jan 16. PMID 19175433
- [Background] Chittock J, Brown K, Cork MJ, Danby SG. Comparing the Effect of a Twice-weekly Tacrolimus and Betamethasone Valerate Dose on the Subclinical Epidermal Barrier Defect in Atopic Dermatitis. Acta Derm Venereol. 2015 Jul;95(6):653-8. doi: 10.2340/00015555-2048. PMID 25594610
- [Background] Chittock J, Cooke A, Lavender T, Brown K, Wigley A, Victor S, Cork MJ, Danby SG. Development of stratum corneum chymotrypsin-like protease activity and natural moisturizing factors from birth to 4 weeks of age compared with adults. Br J Dermatol. 2016 Oct;175(4):713-20. doi: 10.1111/bjd.14568. Epub 2016 Jul 22. PMID 26994359
- [Background] Danby SG, Al-Enezi T, Sultan A, Chittock J, Kennedy K, Cork MJ. The effect of aqueous cream BP on the skin barrier in volunteers with a previous history of atopic dermatitis. Br J Dermatol. 2011 Aug;165(2):329-34. doi: 10.1111/j.1365-2133.2011.10395.x. Epub 2011 Jul 11. PMID 21564067
- [Background] Danby SG, AlEnezi T, Sultan A, Lavender T, Chittock J, Brown K, Cork MJ. Effect of olive and sunflower seed oil on the adult skin barrier: implications for neonatal skin care. Pediatr Dermatol. 2013 Jan-Feb;30(1):42-50. doi: 10.1111/j.1525-1470.2012.01865.x. Epub 2012 Sep 20. PMID 22995032
- [Background] Danby SG, Brown K, Higgs-Bayliss T, Chittock J, Albenali L, Cork MJ. The Effect of an Emollient Containing Urea, Ceramide NP, and Lactate on Skin Barrier Structure and Function in Older People with Dry Skin. Skin Pharmacol Physiol. 2016;29(3):135-47. doi: 10.1159/000445955. Epub 2016 Jun 2. PMID 27251427
- [Background] Danby SG, Chittock J, Brown K, Albenali LH, Cork MJ. The effect of tacrolimus compared with betamethasone valerate on the skin barrier in volunteers with quiescent atopic dermatitis. Br J Dermatol. 2014 Apr;170(4):914-21. doi: 10.1111/bjd.12778. PMID 24328907
- [Background] Petersen LJ. Direct comparison of laser Doppler flowmetry and laser Doppler imaging for assessment of experimentally-induced inflammation in human skin. Inflamm Res. 2013 Dec;62(12):1073-8. doi: 10.1007/s00011-013-0668-2. Epub 2013 Oct 10. PMID 24114290
- [Background] Lu Z, Kasaragod D, Matcher SJ. Conical scan polarization-sensitive optical coherence tomography. Biomed Opt Express. 2014 Feb 18;5(3):752-62. doi: 10.1364/BOE.5.000752. eCollection 2014 Mar 1. PMID 24688811
- [Background] Boncheva M, Damien F, Normand V. Molecular organization of the lipid matrix in intact Stratum corneum using ATR-FTIR spectroscopy. Biochim Biophys Acta. 2008 May;1778(5):1344-55. doi: 10.1016/j.bbamem.2008.01.022. Epub 2008 Feb 11. PMID 18298945
- [Background] Brancaleon L, Bamberg MP, Sakamaki T, Kollias N. Attenuated total reflection-Fourier transform infrared spectroscopy as a possible method to investigate biophysical parameters of stratum corneum in vivo. J Invest Dermatol. 2001 Mar;116(3):380-6. doi: 10.1046/j.1523-1747.2001.01262.x. PMID 11231311
- [Background] Damien F, Boncheva M. The extent of orthorhombic lipid phases in the stratum corneum determines the barrier efficiency of human skin in vivo. J Invest Dermatol. 2010 Feb;130(2):611-4. doi: 10.1038/jid.2009.272. Epub 2009 Sep 3. No abstract available. PMID 19727117
- [Background] Ring A, Schreiner V, Wenck H, Wittern KP, Kupper L, Keyhani R. Mid-infrared spectroscopy on skin using a silver halide fibre probe in vivo. Skin Res Technol. 2006 Feb;12(1):18-23. doi: 10.1111/j.0909-725X.2006.00130.x. PMID 16420534
- [Background] Cooke A, Cork MJ, Victor S, Campbell M, Danby S, Chittock J, Lavender T. Olive Oil, Sunflower Oil or no Oil for Baby Dry Skin or Massage: A Pilot, Assessor-blinded, Randomized Controlled Trial (the Oil in Baby SkincaRE [OBSeRvE] Study). Acta Derm Venereol. 2016 Mar;96(3):323-30. doi: 10.2340/00015555-2279. PMID 26551528
- [Background] Kao JS, Fluhr JW, Man MQ, Fowler AJ, Hachem JP, Crumrine D, Ahn SK, Brown BE, Elias PM, Feingold KR. Short-term glucocorticoid treatment compromises both permeability barrier homeostasis and stratum corneum integrity: inhibition of epidermal lipid synthesis accounts for functional abnormalities. J Invest Dermatol. 2003 Mar;120(3):456-64. doi: 10.1046/j.1523-1747.2003.12053.x. PMID 12603860
- See also: J. Ring, B. Przybilla, and T. Ruzicka, Handbook of Atopic Eczema, J. Ring, B. Przybilla, and T. Ruzicka, Eds., Springer-Verlag, Berlin/Heidelberg (2006) [doi:10.1007/3-540-29856-8] — https://link.springer.com/book/10.1007/3-540-29856-8
- See also: J. Ring, "General Introduction and Epidemiology," in Atopic Dermatitis, pp. 1-25, Springer International Publishing, Cham (2016) [doi:10.1007/978-3-319-22243-1_1]. — https://books.google.co.uk/books?id=DsGuCwAAQBAJ&pg=PA1&lpg=PA1&dq=doi:10.1007/978-3-319-22243-1_1&source=bl&ots=40Co1SDx2v&sig=ACfU3U0oCisZWrOk3VbYMXkSNgLl8ScFNQ&hl=en&sa=X&ved=2ahUKEwjK64yGxuLnAhWUQUEAHeW4AigQ6AEwC3oECAQQAQ#v=onepage&q=doi%3A10.1007%2F978-3-319-22243-1_1&f=false
- See also: Lu, Boadi et al., "Optical coherence tomography demonstrates differential epidermal thinning of human forearm volar skin after 2 weeks application of a topical corticosteroid vs a non- steroidal anti-inflammatory alternative," 85650C (2013) [doi:10.111 — https://www.spiedigitallibrary.org/conference-proceedings-of-spie/8565/1/Optical-coherence-tomography-demonstrates-differential-epidermalthinning-of-human-forearm-volar/10.1117/12.2006104.full?SSO=1